CLINICAL TRIAL: NCT04450316
Title: Low-dose Naltrexone for Bladder Pain Syndrome: A Randomized Placebo-controlled Prospective Pilot Trial
Brief Title: Low-dose Naltrexone for Bladder Pain Syndrome
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study temporarily suspended awaiting research personnel to resume recruitment
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Hah, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 57305
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Bladder Pain Syndrome; Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized on a 1:1 ratio to either LDN or placebo. The randomization sequence will be logged by the study coordinator in a REDCap randomization log blinded to other research staff and clinical team and outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose naltrexone (Active Comparator): 4.5mg of naltrexone to be taken one hour prior to bedtime nightly for 8 weeks.
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): Placebo tablet (sugar-pill) to be taken one hour prior to bedtime nightly for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — 4.5mg tab (low-dose) nightly
  Arms: Low-dose naltrexone
Drug: Placebo — 1 tab nightly
  Arms: Placebo

SUMMARY:
Interstitial cystitis/Bladder Pain Syndrome (IC/PBS) is a constellation of symptoms of pelvic discomfort that includes both bladder-related pain as well as urinary frequency, urgency, and nocturia in the absence of an identifiable etiology that affects likely more than 5.4 million patients in the United States. There is a significant overlap in patients with IC/PBS and those with fibromyalgia and chronic pelvic pain syndrome. Low-dose naltrexone (LDN) has been shown to be effective for the treatment of chronic pain conditions.

The primary aim of this study is to evaluate if LDN improves pain scores and lower urinary tract symptoms in patients with IC/PBS. A secondary aim is to show that it has a low adverse event profile.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with non-Hunner and Hunner lesion disease
* Meeting AUA definition of BPS: An unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder associated with lower urinary tract symptoms of greater than 6 weeks duration in the absence of infection or other identifiable cause.
* Stable treatment for 1 month
* 7-day maximum of pain scores at least 4/10 on the numerical rating scale of pain in the bladder/pelvic area. Urinary frequency 8 or higher while awake. Nocturia 2 or higher. BPIC-SS 19.
* Agreement to not take opioids through the duration of the trial

Exclusion Criteria:

* Substance Use Disorder Diagnosis including Opioid Use Disorder Diagnosis
* Known allergy to naltrexone or naloxone
* Participation in another clinical trial
* Current or planned pregnancy, or breastfeeding
* Chronic pain in another location of the body that is more severe than that related to BPS.
* Any intravesical instillation in last 8 weeks
* If on Elmiron, stable dose for last 3 months
* If on amitriptyline, stable dose for last 3 months
* Any botox within last 6 months
* Treatment for Hunners in the last 6 months
* Any new Interstim settings within last 3 months
* Any new pelvic floor physical therapy in last 12 weeks
* Any change in or new OTC meds over last 2 months.
* Any pain interventions in the preceding 6 weeks (epidural steroid injection, sympathetic block, peripheral nerve block, lumbar medial branch blocks)
* Opioids chronically for IC/BPS in the past unless have been off for 1 year
* Recent short-term (within one week of enrollment) opioid use for flairs
* No documented cystoscopy in the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects in the LDN and placebo groups that are responders with greater than 20% reductions in 7-day average of worst daily Numeric Rating Scale of Pain scores after 8 weeks of treatment. | Will compare pre-intervention to week 8.

SECONDARY OUTCOMES:
Change in Brief Pain Inventory Score | At pre-intervention to week 8.
Change in average frequency and nocturia during a 5-day voiding diary | At pre-intervention to week 8.
Change in Bladder Pain/Interstitial Cystitis Symptom Score | At pre-intervention to week 8
Change in O'Leary Sant symptom scores | At pre-intervention to week 8
Change in O'Leary Sant Problem Indices scores | At pre-intervention to week 8
Change in Global response assessment scale score | At pre-intervention to week 8
Change in PROMIS pain behavior score | At pre-intervention to week 8
Change in PROMIS physical function score | At pre-intervention to week 8
Change in PROMIS sleep dysfunction score | At pre-intervention to week 8
Change in PROMIS Sleep-Related Impairment | At pre-intervention to week 8
Change in PROMIS pain interference score | At pre-intervention to week 8
Change in PROMIS fatigue score | At pre-intervention to week 8
Change in PROMIS anxiety score | At pre-intervention to week 8
Change in PROMIS depression score | At pre-intervention to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Craig V Comiter, MD, Principal Investigator — Stanford University; Phil Hanno, MD, Principal Investigator — Stanford University; Jennifer M Hah, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Should the study result be positive or promising, we would undertake a larger trial at which point we can reassess the sharing of IPD.

REFERENCES:
- [Background] Younger J, Parkitny L, McLain D. The use of low-dose naltrexone (LDN) as a novel anti-inflammatory treatment for chronic pain. Clin Rheumatol. 2014 Apr;33(4):451-9. doi: 10.1007/s10067-014-2517-2. Epub 2014 Feb 15. PMID 24526250